CLINICAL TRIAL: NCT04136197
Title: The Determination of the Trigger Point Incidence After Lumbar Disc Herniation Surgery
Brief Title: Trigger Point Incidence After Lumbar Disc Herniation Surgery
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Ebru Kaya Mutlu, PT, Associate Prof. Dr, PhD, Istanbul University - Cerrahpasa
Other Study IDs: Istanbul University-Cerrahpasa
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Trigger Point Pain, Myofascial
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Manual palpation for incidence determination — The patients are positioned in a sitting and prone lying posture. Trigger points are discrete, local, hypersensitive spots located in a taut band of muscles. Palpation of the trigger point will cause elicitation pain over the affected area and radiation of pain toward a zone of reference and a local twitch response.

SUMMARY:
Our purpose is to determine the incidence of trigger points in patients who remain in a fixed position for a long time during lumbar disc herniation surgery.

DETAILED DESCRIPTION:
The 110 participants between 30-70 years are chosen from patients who had lumbar disc herniation surgery. The trigger points are determined by manually palpating quadratus lumborum, iliocostalis lumborum, gluteus Maximus, gluteus minimus, gluteus medius, ve piriformis muscles before and after surgery. Data will be recorded on the patient assessment file and transferred to the computer and analyzed. Data analysis will be performed with SPSS.20.

ELIGIBILITY:
Inclusion Criteria:

* To be between 30-70 years
* To have low back pain during minimum 6 weeks
* To be voluntary participation for this study
* To approve the informed consent form
* To have the trigger point causing low back pain on muscles including quadratus lumborum, iliocostalis lumborum, gluteus maximus, gluteus minimus, gluteus medius, ve piriformis muscles.

Exclusion Criteria:

* To be diagnosed with spinal stenosis or spondylolisthesis
* To have any skin problem affecting lower extremity evaluation
* To have tumor on spinal region
* To have rheumatological or any systemic problem that may interfere with trigger point diagnose

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients having lumbar disc herniation surgery
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2020-07-18 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Manual Palpation | Change from baseline (preoperative state) to postoperative first and third day
  The patients are positioned in a sitting and prone lying posture.Trigger points are discrete, local, hypersensitive spots located in a taut band of muscles. Palpation of the trigger point will cause elicitation pain over the affected area and radiation of pain toward a zone of reference and a local twitch response.
Visual Analog Scale | Change from baseline (preoperative state) to postoperative first and third day
  Pain will be assessed with Visual Analog Scale (VAS).The VAS is usually a horizontal line, 10 cm in length, anchored by word descriptors at each end with "No Pain" (score of zero) on the left side up to "pain as bad as it could be" or the "worst imaginable pain" (Score of 100 [100-mm scale]) on the right side.The patient was asked to mark the line point that represented his or her current pain.

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Amir Rashedi Bonab, MSc., Study Director — Bahçeşehir University
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kadi F, Waling K, Ahlgren C, Sundelin G, Holmner S, Butler-Browne GS, Thornell LE. Pathological mechanisms implicated in localized female trapezius myalgia. Pain. 1998 Dec;78(3):191-196. doi: 10.1016/S0304-3959(98)00126-2. PMID 9870572
- See also: Pathological mechanisms implicated in localized female trapezius myalgia. — https://www.ncbi.nlm.nih.gov/pubmed/9870572